CLINICAL TRIAL: NCT02570412
Title: Compassionate Use of Aldoxorubicin in Sarcoma Patients Who Have Failed Prior Chemotherapy
Brief Title: Compassionate Use of Aldoxorubicin in Sarcoma Patients Chemotherapy
Status: No longer available | Type: Expanded Access
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Other Study IDs: Aldox Compassionate Use
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — DOXO-EMCH

INTERVENTIONS:
Drug: aldoxorubicin — aldoxorubicin administered at 350 mg/m2

SUMMARY:
Compassionate use of aldoxorubicin in sarcoma patients who have failed prior chemotherapy.

DETAILED DESCRIPTION:
This is a compassionate use protocol allowing sarcoma patients that have relapsed after prior therapies and are not eligible for other protocols involving the evaluation of aldoxorubicin to receive aldoxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unrectable sarcoma that has either relapsed or was refractory to at leat 1 prior chemotherapy or immunotherapy regimen and for which no standard approved therapy exists
* Must not be eligible for another CytRx-sponsored clinical trial
* Able to provide complete medical records for review by the CytRx Medical Monitor
* Able to receive treatment at a site that is participating or has participated in another CytRx-sponsored aldoxorubicin trial
* Capable of providing informed consent and complying with trial procedures
* ECOG performance status 0-2
* Measurable or evaluable tumor lesions according to RECIST 1.1 criteria
* Women must not be able to become pregnant (eg post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study
* Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating

Exclusion Criteria:

* Chemotherapy, palliative surgery and/or radiation treatment less than 30 days prior to screening for non-target lesion
* Exposure to any investigational agent within 30 days of screening
* Central nervous system metastases that are symptomatic
* Laboratory values: Screening serum creatinine >1.5×ULN, ALT >3×ULN, or >5×ULN if liver metastases are present, total bilirubin >3×ULN, ANC <1,500/mm3, platelet concentration <100,000/mm3, hematocrit level <25% for females or <27% for males, coagulation tests (PT, PTT, INR) >1.5×ULN
* Anion gap > 16 meq/L or arterial or venous blood pH < 7.30.
* Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines
* Current serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V
* Baseline QTc >470 msec and/or previous history of QT prolongation while taking other medications. Concomitant use of medications associated with a high incidence of QT prolongation is not allowed
* History or signs of active coronary artery disease with or without angina pectoris.
* Serious myocardial dysfunction defined scintigraphically (eg MUGA, myocardial scintigram) or ultrasound determined absolute LVEF <45% of predicted
* History of HIV infection
* Active, clinically signifiant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals
* Major surgery within 3 weeks prior to enrollment
* Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States